CLINICAL TRIAL: NCT02838108
Title: MURDOCK COPD Observational Study: The Relationship Between GOLD Risk Group and Clinical Outcomes in a Community-based COPD Cohort
Brief Title: The Relationship Between GOLD Risk Group and Clinical Outcomes in a Community-based COPD Cohort
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision to Stop Recruitment
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00072667
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with COPD

SUMMARY:
This is an observational study examining outcomes and treatment patterns in a community-based cohort of subjects with Chronic obstructive pulmonary disease (COPD) who are based in the Kannapolis, NC area.

DETAILED DESCRIPTION:
This study is designed to collect information on the current level of symptoms and ability to breathe, treatment and outcomes of patients with 1) Chronic Obstructive Pulmonary Disease (COPD), or 2) in current or former smokers with respiratory symptoms but preserved pulmonary function or 3) in current or former smokers with respiratory symptoms and preserved ratio with impaired spirometry. This information will be used by the researchers to better understand the impact of COPD on patients. It will also help the researchers study the current recommendations for treatment of COPD.

Chronic obstructive pulmonary disease (COPD) represents a growing public health problem and is now the third leading cause of death in the United States. The risk of exacerbations, hospitalizations and death in patients with COPD tends to increase with increasing severity of airflow limitation. However, the correlation between forced expiratory volume in 1 second (FEV1), symptoms, and health-related quality of life is weak. The shortcomings of using airflow limitation alone to assess the clinical severity of COPD led the Global Initiative for Chronic Obstructive Lung Disease (GOLD) committee to develop a potentially more clinically meaningful approach to assess the impact of COPD on the patient. The GOLD committee has subsequently proposed a model for pharmacologic therapy of patients with stable COPD (i.e. those not currently experiencing a COPD exacerbation) according to GOLD risk group. The therapeutic recommendations proposed by GOLD are widely cited as a strategy for selecting therapy even though this model is predominantly based on expert opinion.

This study will acquire data in a community-based cohort in which patients with COPD or current or former smokers with respiratory symptoms will be classified into GOLD risk groups A-D at enrollment and followed longitudinally. This study will assess the frequency of change in GOLD risk group during 5 years of follow-up, look at the use of COPD medications this cohort and how provider-selected therapy for COPD compares to GOLD-recommended pharmacologic therapy thus addressing a critical knowledge gap in the scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of data collection
* Subjects must be ≥40 years of age
* Subjects must have a greater than or equal to 10 pack-year history of tobacco exposure
* Subjects must have:

  1. COPD confirmed by spirometry performed at screening (as demonstrated by FEV1/FVC < 0.70) or
  2. If the FEV1/FVC is ≥ 0.7, the subject must be a symptomatic current or past Smoker with Respiratory Symptoms (SRS) as defined by meeting the following spirometry and respiratory symptom criteria at screening: FVC ≥ 80% of predicted and CAT score ≥ 10 or
  3. Preserved Ratio Impaired Spirometry (PRISm), defined as a reduced

FEV1 in the setting of a preserved FEV1/FVC ratio:

FEV1/FVC ≥ 0.7 AND FEV1 < 80% of predicted

Exclusion Criteria:

* Participation in an investigational drug trial at the time of screening
* Subjects listed for lung transplantation at the time of screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in The MURDOCK Registry and Biorepository Study cohort who are confirmed to have COPD or are symptomatic current or former smokers.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Composite Endpoint | Measured at the completion of each year of follow-up (years 1, 2, 3, 4 and 5)
  Composite of COPD exacerbation, all-cause hospitalization, and all-cause mortality

SECONDARY OUTCOMES:
Change in COPD Exacerbation | Measured at the completion of each year of follow-up (years 1, 2, 3, 4 and 5)
Change in All-Cause Hospitalization | Measured at the completion of each year of follow-up (years 1, 2, 3, 4 and 5)
Change in Respiratory-related Hospitalization | Measured at the completion of each year of follow-up (years 1, 2, 3, 4 and 5)
Change in All-Cause Mortality | Measured at the completion of each year of follow-up (years 1, 2, 3, 4 and 5)

CONTACTS AND LOCATIONS:
Locations (1):
- MURDOCK Study Office, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoyert DL, Xu J. Deaths: preliminary data for 2011. Natl Vital Stat Rep. 2012 Oct 10;61(6):1-51. PMID 24984457
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Agusti A, Edwards LD, Celli B, Macnee W, Calverley PM, Mullerova H, Lomas DA, Wouters E, Bakke P, Rennard S, Crim C, Miller BE, Coxson HO, Yates JC, Tal-Singer R, Vestbo J; ECLIPSE Investigators. Characteristics, stability and outcomes of the 2011 GOLD COPD groups in the ECLIPSE cohort. Eur Respir J. 2013 Sep;42(3):636-46. doi: 10.1183/09031936.00195212. Epub 2013 Jun 13. PMID 23766334
- [Background] Han MK, Muellerova H, Curran-Everett D, Dransfield MT, Washko GR, Regan EA, Bowler RP, Beaty TH, Hokanson JE, Lynch DA, Jones PW, Anzueto A, Martinez FJ, Crapo JD, Silverman EK, Make BJ. GOLD 2011 disease severity classification in COPDGene: a prospective cohort study. Lancet Respir Med. 2013 Mar;1(1):43-50. doi: 10.1016/S2213-2600(12)70044-9. Epub 2012 Sep 3. PMID 24321803
- [Background] Lange P, Marott JL, Vestbo J, Olsen KR, Ingebrigtsen TS, Dahl M, Nordestgaard BG. Prediction of the clinical course of chronic obstructive pulmonary disease, using the new GOLD classification: a study of the general population. Am J Respir Crit Care Med. 2012 Nov 15;186(10):975-81. doi: 10.1164/rccm.201207-1299OC. Epub 2012 Sep 20. PMID 22997207
- [Background] Soriano JB, Alfageme I, Almagro P, Casanova C, Esteban C, Soler-Cataluna JJ, de Torres JP, Martinez-Camblor P, Miravitlles M, Celli BR, Marin JM. Distribution and prognostic validity of the new Global Initiative for Chronic Obstructive Lung Disease grading classification. Chest. 2013 Mar;143(3):694-702. doi: 10.1378/chest.12-1053. PMID 23187891
- [Background] Centers for Disease Control and Prevention (CDC). Chronic obstructive pulmonary disease among adults--United States, 2011. MMWR Morb Mortal Wkly Rep. 2012 Nov 23;61(46):938-43. PMID 23169314
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Zou H, Hastie T. Regularization and variable selection via the elastic net. Journal of the Royal Statistical Society 2005;series B:301-320.
- [Background] Hans C, Dobra A, West M. Shotgun Stochastic Search for "Large p" regression" Journal of the American Statistical Society 2007;102:507-516.
- [Background] Powell T, Bagnell M. Your "Survival" guide to using time-dependent covariates. SAS Global Forum 2012:68-178.
- [Background] Lin G, So Y, Johnston G. Analyzing survival data with competing risks using SAS system. SAS Global Forum 2012:344-352
- [Background] Elashoff RM, Li G, Li N. A joint model for longitudinal measurements and survival data in the presence of multiple failure types. Biometrics. 2008 Sep;64(3):762-771. doi: 10.1111/j.1541-0420.2007.00952.x. Epub 2007 Dec 20. PMID 18162112